CLINICAL TRIAL: NCT03455595
Title: CONECCT Score so as to Improve the Diagnosis and the Treatment of Colorectal Neoplasia
Brief Title: CONECCT (Colorectal Neoplasia Endoscopic Classification To Chose the Endoscopic Treatment)
Status: Completed | Type: Observational
Sponsor: Hôpital Edouard Herriot (Other)
Responsible Party: Principal Investigator, Jean Christophe Saurin, Professor, Hôpital Edouard Herriot
Other Study IDs: CONECCT
Record Dates: First submitted 2018-02-28; First posted 2018-03-06 (Actual); Last update posted 2018-03-12 (Actual); Status verified 2018-02

CONDITIONS: Digestive System Disease
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic exams — Coloscopy

SUMMARY:
Prospective study so as to evaluate CONECCT score to determine both histological tissue and therapeutic choice

ELIGIBILITY:
Inclusion Criteria:

* N/A

Exclusion Criteria:

* N/A

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Population with colorectal polyps
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the CONECCT endoscopic score so as to improve colon therapeutic treatment polyps | one year
  There are recognized diagnostic criteria so as to predict the histology of colorectal lesions and thus to choose the right therapy. For the moment, these criteria are scattered in at least 5 different classifications and the CONECCT tool will allow gastroenterology interns to more easily predict the histology of the lesion and so to improve the management of them.

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot Hospital, Lyon, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No